CLINICAL TRIAL: NCT02850276
Title: Autonomic Neuropathy, Gastrointestinal Motility, and Inflammation in HIV
Brief Title: Autonomic Neuropathy, GI Motility, and Inflammation in HIV
Acronym: ANGI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Robinson-Papp, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1454; 1R21DK105917-01A1 (NIH)
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: HIV Disease
Keywords: HIV disease; gastrointestinal problems
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyridostigmine (Experimental): 30mg PO three times a day
  Interventions: Drug: Pyridostigmine

INTERVENTIONS:
Drug: Pyridostigmine
  Other Names: Pyridostigmine Bromide; Mestinon; Regonol; Gravitor

SUMMARY:
The purpose of this study is to explore a possible link between the autonomic nervous system and immune function in patients with HIV. Sometimes HIV can cause these nerves to function abnormally, this is called HIV-associated autonomic neuropathy (HIV-AN). HIV-AN is a condition that is different from person to person. In some people it causes no symptoms and is not harmful, in others it may cause symptoms such as dizziness or lightheadedness, nausea, vomiting, diarrhea, constipation, or problems urinating. Most people with HIV-AN don't know that they have it. One of the important nerves in the autonomic nervous system is the vagus nerve. Abnormal function of the vagus nerve may cause stomach and intestinal slowing, which could lead to an overgrowth of bacteria. The body senses these bacteria and tries to fight them, leading to inflammation.

In this study the researchers will test whether abnormal function of the vagus nerve in HIV is associated with stomach slowing and overgrowth of bacteria, and if a drug called pyridostigmine can help.

DETAILED DESCRIPTION:
HIV-infected patients commonly develop autonomic neuropathy (HIV-AN), which is a heterogeneous disorder characterized by varying degrees of both sympathetic and vagal dysfunction. We hypothesize that the vagal component of HIV-AN contributes to chronic inflammation, both directly via loss of cholinergic activity, and indirectly via effects on the GI tract, and that these effects will be treatable using the acetylcholinesterase inhibitor pyridostigmine. The autonomic nervous system controls the inflammatory response to lipopolysaccharide (LPS) via the cholinergic anti-inflammatory pathway. This pathway is mediated by the vagus nerve, and is therefore likely impaired in HIV-AN with vagal dysfunction. Vagal dysfunction also causes slowed GI transit, which could exacerbate LPS-driven inflammation by promoting bacterial overgrowth. However, the anti-inflammatory impact of cholinergic pathways is almost completely unstudied in HIV, despite the known importance of inflammation in HIV disease progression. Therefore, in this exploratory pilot, we seek to establish associations between vagal dysfunction, GI motility and inflammation in virally suppressed, CART-treated individuals with HIV-AN.

Specific Aim 1: To determine whether vagal dysfunction is associated with immune activation in CART-treated participants with HIV-AN, and if so to estimate the extent to which this association is mediated by GI effects (i.e. slowed motility, bacterial overgrowth, microbial translocation) versus direct effects of vagal dysfunction.

Specific Aim 2: In a subset of participants who have both vagal and GI dysfunction, to investigate whether 8 weeks of pyridostigmine: a) reduces immune activation, and b) improves GI motility; and if the immune effect depends on the GI effect.

To achieve these aims, participants with HIV-AN and GI symptoms will be assessed for: vagal dysfunction (heart rate variability); GI dysmotility (gastric emptying scintigraphy); small intestinal bacterial overgrowth (breath testing); microbial translocation (LPS and sCD14); and immune activation (IL-6 and CRP). Participants meeting threshold criteria for both vagal and GI dysfunction will then be treated with pyridostigmine for 8 weeks, after which GI and immune measures will be reassessed.

Objectives Specific Aim 1: To determine whether vagal dysfunction is associated with immune activation in HIV-infected participants treated with combination antiretroviral therapy (CART), and if so to estimate the extent to which this association is mediated by GI effects (i.e. slowed motility, bacterial overgrowth, microbial translocation) versus direct effects of vagal dysfunction.

Specific Aim 2: In a subset of participants who have both vagal and GI dysfunction, to investigate whether 8 weeks of pyridostigmine: a) reduces immune activation, and b) improves GI motility; and if both effects are present to determine whether the immune effect depends on the GI effect.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Documented evidence of HIV-1 infection
* Stable CART therapy for ≥3 months Most recent HIV-1 viral load ≤100 copies/ml (value must be within the past six months)
* English speaking
* Able to tolerate autonomic testing (e.g. able to stand, able to perform Valsalva maneuver).
* If using nicotine-containing products willing to refrain from use for 24 hours prior to all testing procedures (autonomic reflex screen, breath testing, and gastric emptying)
* ≥1 GI symptom on the Survey of Autonomic Symptoms (SAS)47

Exclusion Criteria:

* Diagnosis known to cause autonomic dysfunction other than HIV (e.g. Parkinson's disease, diabetes)
* Diagnosis known to cause GI dysfunction other than HIV (e.g. peptic ulcer disease, infectious diarrhea)
* Current use of any of the following classes of medications (due to potential for significant autonomic or GI effects, interaction with pyridostigmine, or interference with one or more of the testing procedures) Prokinetics (e.g. metoclopramide) Anti-diarrheals (e.g. loperamide) Antibiotics Mefloquine
* Medical or psychiatric conditions precluding safe participation in study procedures or deemed likely to result in hospitalization during the study period.
* The presence of one or more of the following diagnoses which render the Valsalva maneuver relatively or absolutely contraindicated: uncontrolled glaucoma, aortic stenosis, myocardial infarction in the last 6 months, other retinopathy or unclipped cerebral aneurysm.
* The presence of one or more of the following diagnoses which impede interpretation of autonomic testing: cardiac arrhythmias or pacemakers.
* An allergy to eggs (contraindication to gastric emptying scintigraphy)
* Any of the following laboratory results:

Positive pregnancy test (administered to women of childbearing potential only) Urine toxicology screen positive for stimulants (e.g. amphetamines, cocaine) or opiates/opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-11; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robinson-Papp, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with participants in real time if the tests have any clinical significance.

REFERENCES:
- [Background] Deeks SG, Tracy R, Douek DC. Systemic effects of inflammation on health during chronic HIV infection. Immunity. 2013 Oct 17;39(4):633-45. doi: 10.1016/j.immuni.2013.10.001. PMID 24138880
- [Background] Marchetti G, Cozzi-Lepri A, Merlini E, Bellistri GM, Castagna A, Galli M, Verucchi G, Antinori A, Costantini A, Giacometti A, di Caro A, D'arminio Monforte A; ICONA Foundation Study Group. Microbial translocation predicts disease progression of HIV-infected antiretroviral-naive patients with high CD4+ cell count. AIDS. 2011 Jul 17;25(11):1385-94. doi: 10.1097/QAD.0b013e3283471d10. PMID 21505312
- [Background] Robinson-Papp J, Sharma S, Simpson DM, Morgello S. Autonomic dysfunction is common in HIV and associated with distal symmetric polyneuropathy. J Neurovirol. 2013 Apr;19(2):172-80. doi: 10.1007/s13365-013-0160-3. Epub 2013 Apr 12. PMID 23580249
- [Background] Robinson-Papp J, Sharma SK. Autonomic neuropathy in HIV is unrecognized and associated with medical morbidity. AIDS Patient Care STDS. 2013 Oct;27(10):539-43. doi: 10.1089/apc.2013.0188. Epub 2013 Sep 13. PMID 24032624
- [Background] George NS, Sankineni A, Parkman HP. Small intestinal bacterial overgrowth in gastroparesis. Dig Dis Sci. 2014 Mar;59(3):645-52. doi: 10.1007/s10620-012-2426-7. Epub 2012 Oct 5. PMID 23053897
- See also: Related Info — http://www.ncbi.nlm.nih.gov/sites/myncbi/jessica.robinson-papp.1/bibliograpahy/40777172/public/?sort=date&direction=descending

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from November 2015 to Jan 2018
Groups:
- Pyridostigmine: 30mg PO three times a day for 8 weeks
Period: Overall Study
Arm/Group | Pyridostigmine
Started | 76
Completed | 15
Not Completed | 61
Not completed — screen failure | 43
Not completed — Withdrawal by Subject | 14
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 39
  Hispanic/Latino | 22
  White | 14
  Other | 1
Current CD4+ count [Median (Inter-Quartile Range); unit: cells/mm^3] | 602 [464 to 809]
Nadir CD4+ count [Median (Inter-Quartile Range); unit: cells/mm^3] | 200 [56 to 435]
Duration of know HIV infection [Median (Inter-Quartile Range); unit: years] | 21 [17 to 28]
Early Satiety GI symptom [Count of Participants; unit: Participants] | 43
Post-prandial bloating GI symptom [Count of Participants; unit: Participants] | 55
Nausea [Count of Participants; unit: Participants] | 53
Post-prandial vomiting [Count of Participants; unit: Participants] | 15
Cramping/colicky abdominal pain [Count of Participants; unit: Participants] | 41
Moderate to severe diarrhea [Count of Participants; unit: Participants] | 30
Moderate to severe constipation [Count of Participants; unit: Participants] | 31
Vagal sub-score >=1 [Count of Participants; unit: Participants] — Score from 0-3, with higher score indicating more abnormality
  Participants | 30
Adrenal sub-score >=1 [Count of Participants; unit: Participants] — Score from 0-3, with higher score indicating more abnormality
  Participants | 55
Sudomotor sub-score >=1 [Count of Participants; unit: Participants] — Score from 0-3, with higher score indicating more abnormality
  Participants | 63
Total CASS >=3 [Count of Participants; unit: Participants] — Composite Autonomic Severity Score (CASS) which includes sudomotor, vagal, and adrenergic sub-scores. Total Score from 0-10, with higher score indicating more autonomic impairment
  Participants | 49
Autonomic neuropathy CASS vagal subscore >=1 [Count of Participants; unit: Participants] — Score from 0-3, with higher score indicating more abnormality
  Participants | 30
Autonomic neuropathy BRS-V of <4 [Count of Participants; unit: Participants] — vagal baroreflex sensitivity (BRS-V). The vagal component of the baroreflex (BRS_v) is indexed by the heart period (HP) response to changes in BP and is expressed as the regression slope of heart period over SBP during early phase 2.
  Participants | 33
Autonomic neuropathy CASS >=3 [Count of Participants; unit: Participants] — Autonomic neuropathy Composite Autonomic Severity Score (CASS) total Score from 0-10, with higher score indicating more autonomic neuropathy impairment
  Participants | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Breath Test
Description: Breath Test at week 8 as compared to baseline. Breath test results is the rise in the combined hydrogen and methane during the breath test.
Time Frame: baseline and week 8
Measure: Median (Inter-Quartile Range); unit: ppm
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
ppm
  Baseline | 28 [14 to 50]
  week 8 | 14 [9 to 31]

2. Primary Outcome: Number of Participants With Reduction in Small Intestinal Bacterial Overgrowth (SIBO)
Description: Number of participants with reduction in Small intestinal bacterial overgrowth (SIBO) assessed with breath testing after 8 weeks of treatment.
  The hydrogen breath test for the detection of small intestinal bacterial overgrowth (SIBO), obtained by having participants exhale into a plastic bag. the hydrogen content of the samples is measured using a commercially available analyzer.
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
Participants | 13

3. Secondary Outcome: Mean Percent Retention of Gastric Contents on Gastric Emptying Study
Description: Percent retention of gastric contents on gastric emptying study. GI dysmotility calculated from gastric emptying scintigraphy - measurement of the percent retention of gastric contents at 4 hours.
Time Frame: Baseline and week 8
Measure: Mean (Inter-Quartile Range); unit: percent retention of gastric contents
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
percent retention of gastric contents
  Baseline | 3 [2 to 4]
  week 8 | 2 [2 to 4]

4. Secondary Outcome: Change in sCD14 Level
Description: Change in sCD14 level at week 8 as compared to baseline. sCD14 is a marker of macrophage activation commonly used as an indirect measure of translocation
Time Frame: Baseline and week 8
Measure: Median (Inter-Quartile Range); unit: mean florescence intensity
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
mean florescence intensity
  Baseline | 2573 [1859 to 3063]
  Week 8 | 2095 [1784 to 2584]

5. Secondary Outcome: Change in TNFα Level
Description: TNFα is a pro-inflammatory cytokine which is induced by components of translocating bacteria. Change in TNFα level at week 8 compared to baseline
Time Frame: Baseline and week 8
Measure: Median (Full Range); unit: mean florescence intensity
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
mean florescence intensity
  Baseline | 134.0 [114 to 152]
  week 8 | 117.5 [108 to 136]

6. Secondary Outcome: Change in IL-6 Plasma Level
Description: Change in IL-6 plasma level at week 8 as compared to baseline. Plasma interleukin-6 (IL-6), an important inflammatory mediator which predicts mortality in HIV as well as multiple medical co-morbidities, presumably via inflammatory mechanisms.
Time Frame: Baseline and week 8
Measure: Median (Inter-Quartile Range); unit: mean florescence intensity
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
mean florescence intensity
  Baseline | 30.5 [25 to 36]
  Week 8 | 26.5 [23 to 39]

7. Secondary Outcome: The Composite Autonomic Symptom Score (COMPASS)
Description: The gastrointestinal domain domain score of the COMPASS contains 12 items which reflect gastrointestinal symptoms of autonomic function. It is scored on a total scale of 0-28, with higher numbers reflecting worse symptoms.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
score on a scale
  Baseline | 8 (4)
  Week 8 | 8.6 (4.8)

8. Secondary Outcome: Medical Outcomes Study Questionnaire
Description: Medical Outcomes Study (MOS-HIV) quality of life questionnaire. It is a 35 item questionnaire covering 11 dimensions of health including physical functioning, role functioning, pain, social functioning, emotional well-being, energy/fatigue, cognitive functioning, general health, health distress, overall QOL, and health transition. The total scale ranges from 0-100 with a higher score representing better functioning and well-being.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 15
score on a scale
  Baseline | 66.1 (6.2)
  Week 8 | 65 (7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Pyridostigmine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pyridostigmine (N=15)
Stomach Cramps (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1

LIMITATIONS AND CAVEATS:
Limitations include difficulty with recruitment resulting in small sample size, and lack of placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT02850276/Prot_SAP_000.pdf